CLINICAL TRIAL: NCT06002698
Title: Full Pulpotomy Versus Root Canal Treatment for Teeth With Symptomatic Irreversible Pulpitis: A Clinical Study
Brief Title: Full Pulpotomy Versus Root Canal Treatment for Teeth With Symptomatic Irreversible Pulpitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Dr. Hany Mohamed Aly Ahmed, Associate Professor, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DF RD2309/0068 (L)
Record Dates: First submitted 2023-08-09; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Pulpitis - Irreversible

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Root canal treatment (Control) (Other): The procedure can be carried out in single or two visits. Variations in root canal treatment protocols however will make it difficult to compare with pulpotomy so the aim is to standardize the protocols for the following variables including use of rubber dam, Irrigation protocol with 2-2.5% sodium hypochlorite; working length with combined radiographs and apex locators, automated instrumentation to accompany hand instrumentation and preparation to apical size 2-3 larger than the initial binding file. Canal to be medicated with non-setting calcium hydroxide if done in two visits and root canal filling with gutta percha and traditional sealers (warm or cold lateral condensation) and good coronal seal.
  Interventions: Procedure: Root canal treatment (Control)
- Full pulpotomy (Experimental): The clinical procedure will be completed over one or two visits. Following adequate anesthesia and isolation with rubber dam, access to the pulp will be gained following caries removal to de-roof the pulp chamber and excision of the entire coronal pulp. The pulp chamber is irrigated with 2% sodium hypochlorite solution and the resultant bleeding from the remaining pulp will be controlled with a cotton pellet soaked in 2% sodium hypochlorite solution. Following complete haemostasis, the pulp stump will then be covered with Biodentine (Septodont Ltd., Saint Maur des Fausse ́s, France) and the tooth permanently restored with a restoration if treatment is completed in single visit or temporized with glass ionomer cement for the final restoration to be placed in the 2nd visit if operator opted for 2-visit treatment.
  Interventions: Procedure: Full pulpotomy (Experimental)

INTERVENTIONS:
Procedure: Root canal treatment (Control) — Root canal treatment - Removal of the inflamed pulp tissues from the whole root canals of the tooth.
  Arms: Root canal treatment (Control)
Procedure: Full pulpotomy (Experimental) — Full pulpotomy - Removal of the inflamed coronal pulp tissues from the crown of the tooth.
  Arms: Full pulpotomy

SUMMARY:
Background The European Society of Endodontology (ESE) and the American Association of Endodontists (AAE) position statements on the management of deep caries and exposed pulp recommended adoption and promotion of strategies aimed at preserving the pulp, but also acknowledged the need for well-designed and adequately powered randomised control trials to provide the evidence needed to support vital pulp treatment (VPT) and change clinical practice.

Objectives

1. To undertake a randomised controlled clinical trial comparing full pulpotomy with root canal treatment for mature maxillary and mandibular posterior teeth with signs and symptoms indicative of irreversible pulpitis and normal apical tissues in adults.
2. Undertake a cost-effectiveness analysis to examine the potential long-term costs and benefits of pulpotomy.
3. Undertake a process evaluation to assess the acceptability of the intervention to both dentists and patients, while exploring the barriers and enablers to implementation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 12 years or older (with a mature permanent tooth demonstrating radiographic evidence of a deep caries/restorations and signs/ symptoms indicative of IRP (moderate to severe spontaneous lingering pain). Tooth will be responsive to cold and EPT sensibility testing, restorable and can be adequately isolated during treatment. One posterior tooth (molar or premolar) only per patient.

Exclusion Criteria:

* Teeth with active periodontal disease (pocket depth >5mm); teeth indicated for elective root canal treatment for restorative purposes, teeth with apical periodontitis, patients with complex medical histories that may affect their caries experience and healing ability (immunocompromised, radiotherapy), patients who are unable to consent; history of previous trauma to the tooth, presence of apical radiolucency and patients who are pregnant or breast-feeding. Intraoperatively, any evidence of purulence or excessive bleeding that cannot be controlled with a cotton pellet with 2-4% hypochlorite for 10 minutes will be excluded.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Data | 6 months, 1 year and 2 years
  (1) Clinical data: absence of pain, tenderness to palpation, presence of swelling, presence of sinus tract, pathological mobility, response to sensibility testing. Patient history taking and clinical examination for symptoms and clinical signs of infection such as swelling, and sinus tract will be performed by a blinded dental practitioner.
Radiographic data | 6 months, 1 year and 2 years
  (2) Radiographic data: presence of periapical radiolucency, presence of inter-radicular radiolucency, presence of resorption, presence of calcifications. An independent assessor will assess the radiograph obtained at the 12-month review visit.

SECONDARY OUTCOMES:
Post-operative pain | Day 3 and Day 7
  (1) Postoperative pain will be recorded by patients on day 3 and 7. Pain will be assessed using a numeric rating scale (NRS). NRS is an 11-point numeric scale with 0 representing "no pain" and 10 representing "pain as bad as you can imagine". Patients will be instructed on how to use the NRS-11 at home on days 3 and 7 after the procedure. Patients will be contacted by phone call or text message to collect their responses.
Structural integrity assessment | 6 months, 1 year and 2 years
  (2) Structural integrity of the tooth will be assessed by a blinded dental practitioner at the 12-month visit using World Dental Federation (FDI) criteria
Evidence of further interventions and adverse effects | 6 months, 1 year and 2 years
  Evidence of further interventions and adverse events will be obtained from patient records following the 12-month review visit.
Data for cost effective analysis | Baseline, 6 months, 1 year and 2 years
  Data for cost effective analysis and process evaluation will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Hany Ahmed, PhD, Principal Investigator — University of Malaya
Locations (1):
- Hany Mohamed Aly Ahmed, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the IPD.

REFERENCES:
- [Background] European Society of Endodontology (ESE) developed by:; Duncan HF, Galler KM, Tomson PL, Simon S, El-Karim I, Kundzina R, Krastl G, Dammaschke T, Fransson H, Markvart M, Zehnder M, Bjorndal L. European Society of Endodontology position statement: Management of deep caries and the exposed pulp. Int Endod J. 2019 Jul;52(7):923-934. doi: 10.1111/iej.13080. PMID 30664240
- [Background] AAE Position Statement on Vital Pulp Therapy. J Endod. 2021 Sep;47(9):1340-1344. doi: 10.1016/j.joen.2021.07.015. Epub 2021 Aug 3. No abstract available. PMID 34352305
- [Background] Taha NA, Abuzaid AM, Khader YS. A Randomized Controlled Clinical Trial of Pulpotomy versus Root Canal Therapy in Mature Teeth with Irreversible Pulpitis: Outcome, Quality of Life, and Patients' Satisfaction. J Endod. 2023 Jun;49(6):624-631.e2. doi: 10.1016/j.joen.2023.04.001. Epub 2023 Apr 19. PMID 37080387